CLINICAL TRIAL: NCT05321940
Title: A Pilot Safety Trial of STING-dependent Activators (STAVs) and Stimulated Dendritic Cells for Aggressive Relapsed/Refractory Leukemias
Brief Title: Safety Trial of STING-dependent Activators and Stimulated Dendritic Cells for Aggressive Relapsed/Refractory Leukemias
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator decision
Sponsor: Juan C. Ramos, MD (Other)
Responsible Party: Sponsor-Investigator, Juan C. Ramos, MD, Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200982
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-09

CONDITIONS: Refractory Leukemia; Relapsed Leukemia; Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Adult T-Cell Leukemia/Lymphoma
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination STAVs and DC Vaccine Group (Experimental): Participants will receive STAV-loaded cells for a total of 5 doses on Days 3, 17, 31, 45 and 59. Participants will also receive up to 4 doses of dendritic vaccine on Days 10, 17, 24 and 31.
  Interventions: Biological: STING-Dependent Activators (STAVs) Loaded Autologous Leukemic Cells; Biological: Dendritic Cell Vaccine

INTERVENTIONS:
Biological: STING-Dependent Activators (STAVs) Loaded Autologous Leukemic Cells — Autologous human ultraviolet (UV)-irradiated (dead) leukemia cells loaded with STAVs administered via intravenous injection. Each treatment will administer 5 ml via syringe.
  Other Names: STING (Stimulator of Interferon Genes)-Dependent Activators; STAVs-Loaded Autologous Leukemic Cells; STING-dependent innate immune agonists
Biological: Dendritic Cell Vaccine — 15-20 Million mature dendritic cells per dose administered via intravenous injection.
  Other Names: DC Vaccine

SUMMARY:
The purpose of this research is to investigate whether the combination of STING-dependent Adjuvants (STAVs) and dendritic cell (DC) vaccine therapies will increase the body's ability to fight aggressive relapsed or refractory leukemias.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented adult T-cell leukemia/lymphoma (ATLL), Cluster of Differentiation (CD)34+ acute myelogenous leukemia (AML), or acute lymphoblastic leukemia (B-cell or T-cell ALL). Eligible patients with ATLL must have leukemic involvement (See Appendix K for subtype classification).
2. Must have evidence of persistent refractory disease or progression at the time of screening and documented presence of leukemic cells in peripheral blood by either morphology, histology, or flow cytometry.
3. Must have failed standard induction and salvage therapies available AND be ineligible for allogeneic stem cell transplant ǂ as follows:

   For ATLL, must not have failed standard combination chemotherapy (i.e. doxorubicin or etoposide based regimen), salvage chemotherapy (i.e. ifosfamide + carboplatin + etoposide (ICE), dexamethasone, High-dose Cytarabine (Ara-C) and cisplatin (DHAP), or gemcitabine + oxaliplatin (GEMOX)), brentuximab vedotin if CD30+, interferon based therapy if acute or chronic type, and mogamulizumab provided patient is a suitable candidate for the above therapies ±.

   Relapsed/refractory (R/R) AML is defined as patients ≥ 18 years of age at the time of signing the informed consent form (ICF) who are not eligible to receive further intensive therapy and:
   * Have failed to achieve a complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) after induction plus reinduction with intensive chemotherapy (e.g., anthracycline plus cytarabine or high-dose cytarabine containing regimens) if a suitable candidateǂ or 4 cycles of low-intensity therapy (i.e. azacytidine, or decitabine based regimens) (either 4 cycles of the same regimen or a combination of 2 different regimens) OR
   * Have relapsed from CR or CRi from either intensive or low-intensity therapy. Subjects with second or multiple relapses are also eligible.

   For R/R ALL, the patient must have failed (relapsed or primary refractory) induction chemotherapy with consolidation if a suitable candidate± (i.e. ECOG 2993 or similar regimen). The patient should also have failed blinatumomab if CD19+ B-cell ALL, inotuzumab if CD22+ B-cell ALL, tyrosine kinase inhibitor if bcr-abl+, or salvage chemotherapy if available and if the patient is a suitable candidate± for these therapies.

   ± A suitable candidate is defined by a patient who has no contraindications to the available chemotherapy based on organ function, age, and overall health and performance status as determined by the treating physician.

   ǂ Transplant ineligible patients are defined as those not suitable for potentially curative allogeneic stem cell transplant based on lack of disease control or remission at the time of evaluation, inadequate organ function, age, and overall health and performance status as determined by the treating physician, or patient's refusal to undergo such treatment procedure.
4. Adults (≥ 18 years of age) regardless of their gender and genetic background
5. Karnofsky performance status (KPS) ≥ 50% or Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3. (see Appendix B for definitions).
6. Must have adequate end organ and bone marrow function as defined below:
7. Absolute neutrophil count (ANC)≥ 1,000 cells/mm3 (Exception: Unless cytopenias are secondary to leukemia disease).
8. Platelets (PLT) ≥ 50,000 cells/mm3 (Exception: Unless cytopenias are secondary to leukemia).
9. Hepatic function: transaminase ≤ 2.5 x the institutional upper limit of normal, total bilirubin ≤ 1.5 x institutional upper limit of normal, (Exception: Unless secondary to hepatic infiltration with leukemia).
10. Females of childbearing potential (CBP) must have a negative pregnancy test within one week of enrollment. Women should avoid pregnancy while receiving study treatment. Males and females must agree to use adequate methods of birth control during participation in this trial and for 3 months after completing therapy
11. Patients receiving erythropoietin or granulocyte colony-stimulating factor (G-CSF) from baseline are eligible.
12. Ability to understand and willingness to sign a written informed consent document. Written consent by patient or legal guardian on an institutional review board (IRB)-approved informed consent form prior to any study-specific evaluation. Subject or legal guardian must be capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent.

Exclusion Criteria:

1. Patients who have previously received allogeneic stem cell transplant are ineligible
2. Patients receiving cytotoxic chemotherapy within 14 days or any other investigational biological agents within 7 days prior to initiation of study therapy.
3. Any concomitant participation in other therapeutic trials.
4. All patients will be required to be screened for Hepatitis B and C. Patients with active hepatitis B (HBsAg+ and Immunoglobulin M (IgM)+ for Hepatitis B core antigen) will not be eligible for trial enrollment. Those found to be Immunoglobulin G (IgG)+ for Hepatitis core antigen only may be eligible as long as they are receiving anti-Hepatitis B prophylactic therapy and liver function tests meet criteria listed under 4.1.10 above, and have no evidence of cirrhosis. The exact Hepatitis B therapy will be at the discretion of the infection disease specialist or investigator. Participants who are Hepatitis C antibody positive without a positive Hepatitis C RNA level, will be permitted to enroll in the study provided liver function tests meet criteria listed under 4.1.10 above, and have no evidence of cirrhosis on imaging.
5. HIV infection.
6. Active or latent syphilis.
7. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that are likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment.
8. Patients with known central nervous system (CNS) involvement.
9. Pregnant or breast-feeding women.
10. Concurrent active malignancies, with the exception of in situ carcinoma of the cervix, non-metastatic, non- melanomatous skin cancer, or Kaposi's sarcoma not requiring systemic chemotherapy.
11. Known New York Heart Association (NYHA) Class 3 or 4 heart disease as per Appendix C.
12. Known history of cardiomyopathy with ejection fraction < 45% (or lower limit of institutional normal value) or uncontrolled arrhythmia.
13. Psychological, familial, sociological or geographical conditions likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment
14. Known active deep venous thrombosis (DVT) or pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse events | Up to 12 months
  The incidence of treatment-limiting toxicities (TLTs) and treatment-related adverse events, including serious adverse events, in study participants will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Overall Response (OR) | Up to 12 months
  The percentage of participants achieving clinical overall response (complete response (CR) or partial response (PR)) as best response to protocol therapy will be reported. Response will be assessed on the basis of clinical, radiologic, molecular and pathologic (i.e. bone marrow) criteria.
Percentage of Participants Achieving Clinical Complete Response (CR) | Up to 12 months
  The percentage of participants achieving clinical complete response (CR) as best response to protocol therapy will be reported. Response will be assessed on the basis of clinical, radiologic, molecular and pathologic (i.e. bone marrow) criteria.
Percentage of Participants with AML Achieving Clinical Complete Response rate with Incomplete Hematologic Recovery (CRi) | Up to 12 months
  The percentage of participants with acute myelogenous leukemia (AML) achieving clinical complete response with incomplete hematologic recovery (CRi) as best response to protocol therapy will be reported. Response will be assessed on the basis of clinical, radiologic, molecular and pathologic (i.e. bone marrow) criteria.
Percentage of Participants with Minimal Residual Disease (MRD) | Up to 12 months
  The percentage of participants with minimal residual disease after protocol therapy will be reported. Minimal residual disease (MRD) is defined as the persistence of malignant leukemic cells, as detected by conventional morphologic methods (flow cytometry, polymerase chain reaction (PCR), cytogenetics, fluorescence in situ hybridization (FISH), or next generation sequencing), among participants who meet clinical complete response (CR).
Percentage of Participants Achieving Molecular Complete Response (MCR) | Up to 12 months
  The percentage of participants achieving molecular complete response (MCR) will b reported. MCR is defined as no evidence of disease at any body sites below the threshold of detection by conventional morphologic methods pertinent to each study disease (flow cytometry, PCR, T-cell receptor gene rearrangement, cytogenetics, FISH, or next generation sequencing).
Failure-free survival (FFS) rate | Up to 1 year
  Failure-free survival (FFS) is defined as the time from study treatment initiation until documented disease progression, relapse after response, death (by any cause, in the absence of progression), or censoring. In the failure-free subjects, FFS will be censored at the last documented date of failure-free status. FFS rate will be reported as the percentage of participants without progressive disease after start of treatment.
Overall survival (OS) | Up to 1 year
  Overall survival (OS) is defined as the elapsed time from study treatment initiation to death or date of censoring. Participants alive or those lost to follow-up will be censored at the last date known to be alive. OS rate will be reported as the percentage of participants still alive after start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Ramos, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No